CLINICAL TRIAL: NCT03138915
Title: Development and Validation of a Radiomics Signature for Clinically Significant Portal Hypertension in Cirrhosis (CHESS1701): a Prospective Multicenter Study
Brief Title: Radiomics Signature of Hepatic Venous Pressure Gradient (rHVPG) With CT Angiography (CHESS1701)
Acronym: rHVPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing 302 Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Beijing YouAn Hospital (Other); Xingtai People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, M.D., Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHESS1701
Record Dates: First submitted 2017-04-29; First posted 2017-05-03 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hypertension, Portal
Keywords: clinically significant portal hypertension; hepatic venous pressure gradient; radiomics
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Patients will receive CTA, HVPG measurement, and rHVPG per protocol. Intervention: Procedure: HVPG measurement
  Interventions: Procedure: HVPG measurement; Procedure: CTA

INTERVENTIONS:
Procedure: HVPG measurement — HVPG obtained by means of catheterization of a hepatic vein with a balloon catheter.
Procedure: CTA — Radiomic features were extracted from CTA images.

SUMMARY:
This is a prospective, multi-center diagnostic trial conducted at 5 high-volume liver centers in China designed to determine the diagnostic performance of radiomics-based hepatic venous pressure gradient (rHVPG) (investigational technology) by CT angiography (CTA) for noninvasive assessment of the clinically significant portal hypertension (CSPH) in patients with cirrhosis. Direct hepatic venous pressure gradient (HVPG) measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH, which is defined as HVPG≥10 mmHg.

DETAILED DESCRIPTION:
This is a prospective, multi-center diagnostic trial conducted at 5 high-volume liver centers (302 Hospital of PLA; Beijing Shijitan Hospital; The Third Xiangya Hospital of Central South University; Beijing Youan Hospital; Xingtai People's Hospital) in China designed to determine the diagnostic performance of radiomics-based hepatic venous pressure gradient (rHVPG) (investigational technology) by CT angiography (CTA) for noninvasive assessment of the clinically significant portal hypertension (CSPH) in patients with cirrhosis. Direct hepatic venous pressure gradient (HVPG) measurement by means of catheterization of a hepatic vein with a balloon catheter is the gold-standard method to assess the presence of CSPH, which is defined as HVPG≥10 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients providing written informed consent
* Patients with cirrhosis and scheduled to undergo clinically-indicated invasive HVPG measurement by means of catheterization of a hepatic vein with a balloon catheter
* Has undergone > 64 multi-detector row CT within 14 days prior to hepatic vein catheterization
* No hepatic-portal vein interventional therapy between the CT and hepatic vein catheterization

Exclusion Criteria:

* Prior transjugular intrahepatic portosystem stent-shunt surgery
* Prior devascularization operation
* Has received a liver transplant
* Patients with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status
* Patient requires an emergent procedure
* Any active, serious, life-threatening disease
* Inability to adhere to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-10-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of rHVPG | 1 day
  Diagnostic accuracy of rHVPG to determine presence or absence of a CSPH when compared to HVPG as the reference standard (HVPG≥10mmHg)

SECONDARY OUTCOMES:
Diagnostic Performance of rHVPG | 1 day
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of rHVPG when compared to HVPG as the reference standard (HVPG≥10mmHg)
rHVPG Numerical Correlation | 1 day
  Correlation of the rHVPG numerical value with the HVPG numerical value

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (6):
- China (6):
  - 302 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833
- [Derived] Wang C, Huang Y, Liu C, Liu F, Hu X, Kuang X, An W, Liu C, Liu Y, Liu S, He R, Wang H, Qi X. Diagnosis of Clinically Significant Portal Hypertension Using CT- and MRI-based Vascular Model. Radiology. 2023 Apr;307(2):e221648. doi: 10.1148/radiol.221648. Epub 2023 Jan 31. PMID 36719293
- [Derived] Liu Y, Ning Z, Ormeci N, An W, Yu Q, Han K, Huang Y, Liu D, Liu F, Li Z, Ding H, Luo H, Zuo C, Liu C, Wang J, Zhang C, Ji J, Wang W, Wang Z, Wang W, Yuan M, Li L, Zhao Z, Wang G, Li M, Liu Q, Lei J, Liu C, Tang T, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Ellik Z, Asiller OO, Liu Z, Teng G, Chen Y, Hou J, Li X, He X, Dong J, Tian J, Liang P, Ju S, Zhang Y, Qi X. Deep Convolutional Neural Network-Aided Detection of Portal Hypertension in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2998-3007.e5. doi: 10.1016/j.cgh.2020.03.034. Epub 2020 Mar 21. PMID 32205218